CLINICAL TRIAL: NCT02745197
Title: Factors That Regulate Components of a Nutritional Supplement to Support Skeletal Muscle in Cancer Patients
Brief Title: A Study to See Whether a Nutritional Supplement is Beneficial for Patients With Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: change in concept
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HREBA-CC-15-0218
Record Dates: First submitted 2016-01-13; First posted 2016-04-20 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2018-10

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional Supplement (Experimental): 2 nutritional supplement capsules, taken by mouth 3 times per day, for approximately 10 to 15 weeks.
  Interventions: Dietary Supplement: Nutritional Supplement
- Placebo (Placebo Comparator): 2 placebo capsules, taken by mouth 3 times per day, for approximately 10 to 15 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement — Participants will take 2 capsules, containing the nutritional supplement, 3 times per day.
  Arms: Nutritional Supplement
Dietary Supplement: Placebo — Participants will take 2 capsules, containing a placebo, 3 times per day.
  Arms: Placebo

SUMMARY:
This study evaluates a nutritional supplement in the treatment of pancreatic cancer in adults. Half of the participants will receive the nutritional supplement, while the other half will receive a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a newly diagnosed pancreatic tumor thought to be pancreatic cancer scheduled for resection of the tumor.
* Patients with a newly diagnosed pancreatic tumor thought to be pancreatic cancer, subsequently found to have biliary or ampullary cancer upon full pathological review, scheduled for resection of the tumor.
* Patients with a CT image, which includes scans of the 3rd lumbar region, taken within 45 days before tumor resection surgery.
* Ability to maintain oral intake.
* Ability to give written, informed consent.

Exclusion Criteria:

* Patients found to have a diagnosis other than pancreatic, biliary, or ampullary cancer upon full pathological review.
* Patients with a benign tumor.
* Patients taking drugs that modify muscle metabolism.
* Patients with uncontrolled jaundice.
* A compliance rate of <80%, excluding compliance during recovery from tumor resection surgery while in the hospital.
* Patients currently taking the nutritional supplement being investigated in this study.
* Patients in the placebo group who have plasma levels of the nutritional supplement components within the range of the nutritional supplement group at study time points when plasma levels of the nutritional supplement components are significantly higher in the nutritional supplement group versus the placebo group.
* Inadequate specimens.
* Known allergy to gelatin or glycerin.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Muscle fatty acid content | At time of tumor removal surgery
  Quantification of muscle triglyceride fatty acid (ug/g)

SECONDARY OUTCOMES:
Plasma levels of the nutritional supplement | Baseline (before initiation of capsule consumption), day of tumor removal surgery (an average of 2-5 weeks from baseline), and day of post-surgery follow-up CT scan (an average of 8-10 weeks after surgery)
  Quantification of the plasma concentration of nutritional supplement components (ug/mL)
Determine computed tomography (CT)-derived body composition | Within 45 days before tumor removal surgery, and day of post-surgery follow-up CT scan (an average of 8-10 weeks after surgery)
  Quantitatively determine body composition as assessed by computed tomography (CT) scans, relative to stature (cm2/m2)
Plasma C-reactive protein | Baseline (before initiation of capsule consumption), day of tumor removal surgery (an average of 2-5 weeks from baseline), and day of post-surgery follow-up CT scan (an average of 8-10 weeks after surgery)
  Plasma quantification of C-reactive protein (mg/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Vera Mazurak, Ph.D., Principal Investigator — University of Alberta